## INFORMED CONSENT FORM

| Official Study Title | Comparison of the Effects of Vaginal Cuff<br>Closure Techniques on Vaginal Length and<br>Sexual Function in Laparoscopic<br>Hysterectomy |
|---|---|
| Document Date | 01/05/2022 |

This study you are participating in is a scientific study, and the title is "Comparison of the effects of vaginal vault closure techniques in laparoscopic hysterectomy on vaginal length and sexual life." The purpose of this study was to compare the effects of vaginal vault closure techniques in laparoscopic hysterectomy on vaginal length and women's sexual life. We used the Arizona Sexual Experiences Scale to assess women's sexual life. In this study, you will be examined before surgery and filled out a form. Three months after surgery, you will be called and referred to the Department of Obstetrics and Gynecology for a re-evaluation.

You will not be paid for your participation in this study; furthermore, no fees will be charged to you or your social security institution for all examinations, tests, and medical care services provided within the scope of this study. Participation in this study is entirely voluntary. You may refuse to participate or withdraw from the study at any stage; this will not result in any penalty or hindrance to your benefits. The researcher may remove you from the study, with or without your knowledge, for reasons such as failure to comply with the treatment plan, disruption of the study program, or to enhance the effectiveness of the treatment. The results of the study will be used for scientific purposes; your withdrawal from the study or the researcher's decision to withdraw from the study will be If you are removed, your medical data may also be used for scientific purposes if necessary. All of your medical and identity information will be kept confidential, and your identity will not be disclosed even if the study is published. However, research investigators, investigators, ethics committees, and official authorities may access your medical information if necessary. You may also access your own medical information at any time.

Consent to Participate in the Study: I have read and listened to the information listed above, which must be provided to the subject before the study begins. I have asked the researcher all questions I can think of and have fully understood all the explanations given to me, both verbally and in writing. I have been given sufficient time to decide whether I wish to participate in the study. Under these circumstances, I authorize the researcher to review, transfer, and process my medical information, and I accept the invitation to participate in this study voluntarily, without any coercion or pressure.

I will be provided with a signed copy of this form.